CLINICAL TRIAL: NCT07302334
Title: A Feasibility Study of Group-Based Metacognitive Therapy (MCT) for Post-Traumatic Stress Disorder (PTSD) in a Routine Healthcare Setting
Brief Title: Feasibility of Group-Based Metacognitive Therapy for PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Maria Bragesjo, Prinicipal investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-03111-01
Record Dates: First submitted 2025-11-28; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: PTSD
Keywords: PTSD; MCT
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Meta-cognitive therapy will be offered in a group-based format for 14 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group-based metacognitive therapy (Experimental): 14 weeks of group-based meta-cognitive therapy
  Interventions: Behavioral: Group-based metacognitive therapy

INTERVENTIONS:
Behavioral: Group-based metacognitive therapy — Group-based metacognitive therapy will be offered for 14 weeks.

SUMMARY:
The primary objective of this study is to investigate the feasibility and acceptability of group-based Metacognitive Therapy (MCT) for post-traumatic stress disorder (PTSD) when delivered within routine psychiatric care in Sweden.

The secondary objective is to evaluate preliminary treatment effects of group-based MCT on symptoms of post-traumatic stress, complex PTSD, depression, and quality of life, and to compare treatment dropout rates to those reported in the existing literature on exposure-based treatments for PTSD.

DETAILED DESCRIPTION:
The investigators will investigate a 14 weekly group-based Metacognitive Therapy (MCT) for post-traumatic stress disorder (PTSD). Feasibility and acceptability outcomes include recruitment and retention rates, data completeness, treatment adherence, and qualitative evaluations of patient experiences. Recruitment is designed to be broadly inclusive with minimal exclusion criteria. Patients will be recruited from a psychiatric clinic specialised in PTSD in Stockholm, Sweden. The investigators hypothesize that group-based MCT will result in significant within-group reductions in PTSD and depressive symptoms and improvements in functioning and quality of life from pre- to post-treatment, with effects maintained up to the 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Fulfills the diagnostic criteria for PTSD based on clinical records
* Self-rated total sum score over 30 on the PCL-5
* Age ≥18 years.
* Stable psychotropic medication regimen for ≥4 weeks.
* Fluent in Swedish.

Exclusion Criteria:

* Severe psychiatric comorbidities (e.g., suicidal ideation, active psychosis, bipolar disorder) warranting immediate attention.
* Current trauma-related threat (e.g., ongoing domestic violence).
* Ongoing evidence-based trauma-focused psychological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants that conducts the weekly measures and further assessment points | Through study completion up to the 6 months follow up
  The proportion of participants that conducts the weekly measures and further assessment points
The proportion of participants that go through the entire treatment period | Completion of treatment period, up to the last session delivered 14 weeks after treatment start
  The proportion of participants that go through the entire treatment period
Adverse events related to the treatment | Through study completion, up to the 6 months follow up
  Adverse events related to the treatment
Acceptability | Completion of treatment period, up to the last session delivered 14 weeks after treatment start
  Number of drop-outs from treatment
Treatment acceptability | Baseline
  Number of individuals offered the intervention but declined part of treatment
Treatment acceptability | Up to 6 months after treatment completion
  Participants experience/satisfaction with treatment and assessment procedures through qualitative interviews
Participants satisfaction with treatment, assessed by The Client Satisfaction Questionnaire (CSQ-8). | Up till treatment completion, 14 weeks after treatment start
  The CSQ-8 yields a single score measuring a single dimension of overall satisfaction. An "overall score" is calculated by summing the score on each of the eight scale item. Scores range from 8 to 32, with higher values indicating higher satisfaction.
Treatment adherence | Up to treatment completion, 14 weeks after treatment start.
  The proportion of completed group-sessions

SECONDARY OUTCOMES:
Change in PTSD symptoms as assessed by the PTSD Check List - DSM-5 (PCL-5) | At baseline, after seven weeks of treatment, immediately after treatment completion, at 3-month and 6-months follow up after treatment completion.
  The PCL-5 is a 20-item self-report measure based upon the Diagnostic and Statistical Manual (DSM-5) criteria for PTSD. Total Score (Range 0-80 with higher scores representing more PTSD symptoms.
Change in ICD-11 PTSD and complex PTSD symptoms as assessed by the International Trauma Questionnaire (ITQ). | At baseline, immediately after treatment completion, at 3-month and 6-months follow up after treatment completion.
  The ITQ includes six items measuring each PTSD symptom cluster and these items measure how bothersome each symptom has been in the past month. The ITQ also includes six items measuring each 'Disturbance in Self-Organization' (DSO) symptom in complex PTSD. These items measure how a respondent typically feels, thinks about oneself, and relates to others. The PTSD and DSO symptoms are accompanied by three items measuring associated functional impairments in the domains of social, occupation, and other important areas of life. All items are answered on a 5-point Likert scale ranging from 0 (Not at all) to 4 (Extremely). Thus, PTSD and DSO symptom scores range from 0 to 24 and CPTSD symptom scores range from 0 to 48. Higher scores represents more PTSD and complex PTSD symptoms.
Change in depressive symptoms as measured by the Patient Health Questionnaire-9 (PHQ-9) | At baseline, immediately after treatment completion, at 3-month and 6-months follow up after treatment completion.
  The PHQ-9 is a widely used and well-validated instrument for measuring the severity of depressive symptoms. Scores are calculated based on how frequently a person experiences 9 symptoms of depression ranging from "not at all" response is scored as 0; "several days" response is 1; "more than half the days" response is 2; and "nearly every day" response is 3. Higher scores represents more depressive symptoms.
Change in quality of life measured by Euroqol, EQ-5D | At baseline, immediately after treatment completion, at 3-month and 6-months follow up after treatment completion.
  Change in overall health from baseline to post treatment and follow up . EQ-5D is a standardized self-report measure of overall health status measured in terms of five dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using a three-level scale: 1 having no problems, 2 having some problems and 3 having extreme problems. A higher score indicate worse severity.
Change in tendency to engage in excessive, uncontrollable, and generalized worry measured by PSWQ | At baseline, immediately after treatment completion, at 3-month and 6-months follow up after treatment completion.
  Change in tendency to engage in excessive and uncontrollable worry from baseline to post-treatment and follow-up.
  The Penn State Worry Questionnaire (PSWQ) is a standardized self-report measure assessing the general tendency to experience persistent, excessive, and uncontrollable worry. It measures the extent to which worry is perceived as pervasive, distressing, and difficult to control across situations. The scale consists of 16 items rated on a 5-point Likert scale ranging from 1 ("not at all typical of me") to 5 ("very typical of me"). Items reflect frequency, intensity, and uncontrollability of worry. Higher scores indicate a greater tendency toward pathological worry.
Change in general anxiety level measured by GAD-7 | At baseline, immediately after treatment completion, at 3-month and 6-months follow up after treatment completion.
  Change in The Generalized Anxiety Disorder scale (GAD-7), a standardized self-report measure of general anxiety symptoms. It consists of 7 items assessing the frequency of core anxiety symptoms such as excessive worry, tension, restlessness, irritability, and difficulties relaxing or concentrating. Respondents rate how often they have been bothered by each symptom over the past two weeks on a 4-point scale ranging from 0 ("not at all") to 3 ("nearly every day"). Total scores range from 0 to 21, with higher scores indicating more severe anxiety.
Adverse events related to treatment measured by the Negative effects questionnaire-20. | Immediately after treatment completion, at 3-month and 6-months follow up after treatment completion.
  Self-rated questionnaire on negative effects. It contains 20 items that are scored on a five point Likert-scale (0-4) and differentiates between negative effects that are attributed to treatment and those possibly caused by other circumstances. The total score of the NEQ ranges from 0 to 80 points, a higher score reflects more negative effects.

OTHER OUTCOMES:
Dropout Rates | Immediately after treatment completion
  Drop out rates will be compared with published data on trauma-focused CBT and EMDR for PTSD.

CONTACTS AND LOCATIONS:
Locations (1):
- Affektiva, ångest och traumaprogrammet, Psykiatri Sydväst, Stockholm, Sweden